CLINICAL TRIAL: NCT06506539
Title: Clinical and Laboratory Evaluation of Placenta Extract Gel as an Adjunct to Non Surgical Periodontal Therapy in Patients With Grade B Stage II Periodontitis
Brief Title: Placenta Extract Gel as a Periodontal Local Delivery Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Aya mohamed ahmed awad, dr, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 336/2021
Record Dates: First submitted 2024-07-06; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Pocket; Periodontitis
Keywords: placenta extract gel; periodontitis; local delivery drug
MeSH Terms: conditions — Periodontal Pocket; Periodontitis | interventions — Placental Extracts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling and root planning only (No Intervention)
- scaling and root planning+planenta extract gel group (Active Comparator)
  Interventions: Drug: Placental Extract

INTERVENTIONS:
Drug: Placental Extract — add placental extract gel as a local delivery drug in periodontal pocket
  Arms: scaling and root planning+planenta extract gel group

SUMMARY:
Introduction: Periodontal disease is one of the most prevalent global chronic disorders. Pathology affecting the structure surrounding teeth results in inflammation initiated by bacterial aggregation and alteration in their profile.

conventional periodontal therapeutics has focused on the control of etiologic agents, thereby promoting healing, repair of tissues delivery of therapeutic agents into the pocket act as drug reservoirs which could alter pathogenic flora and promote its repair and wound healing. Aim of the study: Evaluate the effect of locally delivered placenta extract gel as an adjunct to scaling and root planning in the treatment of periodontal pocket. Methodology: 30 patients with grade B stage II periodontitis will be selected from the Faculty of Dentistry Suez Canal University outpatient clinic and divided into 2 equal groups. Group I: will have scaling and root planning.

Group II: will have scaling and root planning with placenta extract gel locally delivered in the periodontal pocket. All clinical parameters (plaque index, gingival index, probing pocket depth, and clinical attachment) and lab investigations (vascular endothelial growth factor and fibroblast growth factor) will be measured at 0,1 and 3 months. All results will be tabulated and statistically analyzed using the SPSS program.

DETAILED DESCRIPTION:
Group I: (control group): where subgingival scaling and root planning will be performed and the pocket will be allowed to heal with secondary intention. Group II (test group): where subgingival scaling and root planing, and 1ml of human placental extracts gel* adsorbed in 30 beads of gelatin foam of 1sq. mm, will be placed into the pockets with the help of a probe to fill the sulcus to the deepest point & coepak will be placed. patients will be recalled after seven 12 days to remove the coePak. A customized acrylic stent will be fabricated for each patient to provide a reproducible insertion axis for the periodontal probe. The stent will be grooved in an occlusal-apical direction for the above-mentioned purpose.

Lab assessment:

The area will be isolated with cotton rolls, gingival crevicular fluid will be collected using a paper point three times for each pocket, and samples will be stored at -80°.

Vascular endothelial growth factor and fibroblast growth factor will be measured for the two groups using the ELISA technique.

Clinical assessment:

The following parameters will be recorded for the two groups: plaque index, gingival index depth, probing pocket, and clinical attachment.(Silness and Löe, 1964, Löe and Silness, 1963) Measurements will be taken from the stent to the deepest probing depth to record. Probing pocket depth (PPD) while Relative Attachment level (RAL) will be recorded by subtracting the length of the deepest probing depth from the stent from the length from the stent to the cemento-enamel junction All the clinical parameters will be recorded on day 0,1 months and 3 months and all results will be tabulated and statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

- having a pocket of 4-5 mm ( grade B stage II periodontitis).

Exclusion Criteria:

* patients with known systemic conditions like Diabetes mellitus, hypertension, atherosclerosis, and other conditions known to affect periodontal status adversely.
* patients suffering from stage III grade C periodontitis.
* pregnant and lactating women,
* known harmful habits like alcohol consumption, and tobacco.
* any form of periodontal therapy during the last six months & antimicrobial therapy during the last 3 months.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
plaque index (PI) | 3 months
  PI was used to determine the amount of plaque on the tooth surface
  To determine the plaque index, Silness & Löe reference values were taken as a basis:
  Plaque index 0: No plaque is in the area adjacent to the gingiva. Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
  Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
  Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.
gingival index (GI) | 3 months
  o determine the gingival index of the patients, gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of all teeth was evaluated. The gingival index of an individual was obtained by summing the values determined for each tooth and calculating the averages. To determine the gingival index, Löe & Silness reference values were taken as a basis: Gingival index 0: Healthy gums. Gingival index 1: Mild discolouration and oedematous gingiva. No bleeding on probing.
  Gingival index 2: Red, oedematous and shiny gingiva. There is bleeding on probing.
  Gingival index 3: Red, oedematous, and ulcerated gingiva. There is spontaneous bleeding.
probing pocket depth (PD) | 3 months
  Measured from the free gingival margin to the bottom of the pocket with an unc 15 periodontal probe
clinical attachment level(CAL). | 3 months
  The distance from CEJ to the bottom of the pocket. It was measured in the same way described for probing depth.
  CAL was recorded by subtracting the length of the deepest probing depth from the stent by the length from the stent to the cemento-enamel junction.

SECONDARY OUTCOMES:
Vascular endothelial growth factor (VEGF) | 3 months
  recorded in picograms per milliliter (pg/mL)
fibroblast growth factor (FGF) | 3 months
  recorded in picograms per milliliter (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: dalia fayad, Phd, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464